CLINICAL TRIAL: NCT01992458
Title: Observatoire Multicentrique Français Des Porteurs de Défibrillateur Automatique Implantable en Prévention Primaire (Cardiopathie Ischémique ou Cardiomyopathie Dilatée)
Brief Title: Primary Prevention ICD French Registry
Acronym: DAI-PP
Status: Completed | Type: Observational
Sponsor: Clinique Pasteur (Other)
Collaborators: Clinique Pasteur Toulouse (Other); European Georges Pompidou Hospital (Other); University Hospital, Grenoble (Other); University Hospital, Bordeaux (Other); University Hospital, Lille (Other); University Hospital, Marseille (Other); Centre Cardiologique du Nord, St Denis (Unknown); Nouvelles Cliniques Nantaises, Nantes (Unknown); Hopital Antoine Beclere, Clamart (Unknown); Rennes University Hospital (Other); Central Hospital, Nancy, France (Other); University Hospital, Tours (Other)
Responsible Party: Principal Investigator, Serge Boveda, MD, Clinique Pasteur
Other Study IDs: 913203
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Evaluation of Primary Prevention ICD in Real Life
Keywords: implantable cardioverter defibrillator; death; shock; mortality; complication; sudden death
MeSH Terms: conditions — Death; Shock; Death, Sudden

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The indication of implantable cardioverter defibrillator (ICD) therapy for primary prevention of sudden cardiac death has been introduced later in France than in other parts of the World. Overall, we aimed to assess the risk-benefit ratio of this strategy over a 10 year period.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease or dilated cardiomyopathy with low ejection fraction implanted with an ICD in the setting of primary prevention (criteria at the discretion of the physician)

Exclusion Criteria:

* Setting of secondary prevention
* Other cardiopathies such as congenital, channelopathies, valvulopathies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients from 12 medical centers implanted with an implantable cardioverter defibrillator (ICD) in the setting of primary prevention since Jan. 1, 1997, in France
Sampling Method: Non-Probability Sample
Enrollment: 5576 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Incidences of Appropriate Therapies (ATP and Shocks) and ICD-Related Complications | 3-year

SECONDARY OUTCOMES:
Cause-of-Death Analysis | 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Serge Boveda, MD, Principal Investigator — Clinique Pasteur; Eloi Marijon, MD, Principal Investigator — Hopital européen Georges Pompidou
Locations (1):
- Clinique Pasteur, Toulouse, France

REFERENCES:
- [Derived] Escande W, Boveda S, Defaye P, Leclercq C, Sadoul N, Perier MC, Deharo JC, Fauchier L, Marijon E, Piot O; DAI-PP Investigators. Outcomes in Guideline-Based Versus Off-Guideline Primary Prevention Implantable Cardioverter-Defibrillator Recipients. J Am Coll Cardiol. 2017 Sep 5;70(10):1302-1303. doi: 10.1016/j.jacc.2017.07.711. No abstract available. PMID 28859794
- [Derived] Amara N, Boveda S, Defaye P, Klug D, Treguer F, Amet D, Perier MC, Gras D, Algalarrondo V, Bouzeman A, Piot O, Deharo JC, Fauchier L, Babuty D, Bordachar P, Sadoul N, Marijon E, Leclercq C; DAI-PP Investigators. Implantable cardioverter-defibrillator therapy among patients with non-ischaemic vs. ischaemic cardiomyopathy for primary prevention of sudden cardiac death. Europace. 2018 Jan 1;20(1):65-72. doi: 10.1093/europace/euw379. PMID 28082419
- [Derived] Clementy N, Challal F, Marijon E, Boveda S, Defaye P, Leclercq C, Deharo JC, Sadoul N, Klug D, Piot O, Gras D, Bordachar P, Algalarrondo V, Fauchier L, Babuty D; DAI-PP Investigators. Very high rate programming in primary prevention patients with reduced ejection fraction implanted with a defibrillator: Results from a large multicenter controlled study. Heart Rhythm. 2017 Feb;14(2):211-217. doi: 10.1016/j.hrthm.2016.10.024. Epub 2016 Oct 28. PMID 27989789
- [Derived] Escande W, Marijon E, Defaye P, Piot O, Leclercq C, Sadoul N, Deharo JC, Empana JP, Boveda S, Klug D. Electrical Storms in Patients With Implantable Cardioverter-Defibrillators for Primary Prevention. J Am Coll Cardiol. 2016 Sep 13;68(11):1248-1250. doi: 10.1016/j.jacc.2016.06.039. No abstract available. PMID 27609689
- [Derived] Providencia R, Marijon E, Lambiase PD, Bouzeman A, Defaye P, Klug D, Amet D, Perier MC, Gras D, Algalarrondo V, Deharo JC, Leclercq C, Fauchier L, Babuty D, Bordachar P, Sadoul N, Piot O, Boveda S. Primary Prevention Implantable Cardioverter Defibrillator (ICD) Therapy in Women-Data From a Multicenter French Registry. J Am Heart Assoc. 2016 Feb 12;5(2):e002756. doi: 10.1161/JAHA.115.002756. PMID 26873687